CLINICAL TRIAL: NCT05047939
Title: Comparison of Recovery Profile After Total Intravenous Anesthesia Between Remimazolam With Flumazenil and Propofol in Patients Undergoing Thyroidectomy: A Single-blinded Randomized Controlled Trial
Brief Title: Comparison of Recovery Profile After TIVA Between Remimazolam With Flumazenil and Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Hana Pharm Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2105-016-1217
Record Dates: First submitted 2021-08-23; First posted 2021-09-17 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia, Intravenous
Keywords: Anesthetics; Anesthetics, General; Benzodiazepines; Flumazenil

STUDY DESIGN:
Intervention Model Description: A prospective randomized single-blinded study
Who Masked: Participant
Masking Description: Patients will receive general anesthesia, therefore they cannot know their anesthetic agents.
  Physicians involved in this study will investigate the outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remimazolam group (Experimental): In the remimazolam-based TIVA group, general anesthesia is induced and maintained with a continuous infusion of remimazolam using an infusion pump. In the remimazolam group, its antagonist, flumazenil 0.2mg, is administered at the end of surgery. In both groups, remifentanil is continuously infused throughout the surgery for balanced anesthesia, adjusted to maintain arterial pressure.
  Interventions: Drug: remimazolam-based TIVA
- propofol group (Active Comparator): In the propofol-based TIVA group, general anesthesia is induced and maintained with a target-controlled infusion of propofol using an infusion pump (Orchestra®; Fresenius Vial, France). In both groups, remifentanil is continuously infused throughout the surgery for balanced anesthesia, adjusted to maintain arterial pressure.
  Interventions: Drug: propofol-based TIVA

INTERVENTIONS:
Drug: remimazolam-based TIVA — In the remimazolam-based TIVA group, general anesthesia is induced and maintained with a continuous infusion of remimazolam using an infusion pump. In the remimazolam group, its antagonist, flumazenil, is administered at the end of surgery.
  Other Names: remimazolam group
  Arms: remimazolam group
Drug: propofol-based TIVA — In the propofol-based TIVA group, general anesthesia is induced and maintained with a target-controlled infusion of propofol using an infusion pump (Orchestra®; Fresenius Vial, France).
  Other Names: propofol group
  Arms: propofol group

SUMMARY:
This prospective, randomized, single-blinded study is designed to compare the recovery profile between propofol-based total intravenous anesthesia (TIVA) and remimazolam-based TIVA in patients undergoing thyroidectomy. In the remimazolam group, its antagonist, flumazenil, is administered at the end of surgery. We hypothesize that remimazolam-based TIVA antagonized by flumazenil can significantly shorten the time from the end of anesthetic administration to eye-opening compared to propofol-based TIVA.

DETAILED DESCRIPTION:
Adult patients undergoing elective thyroidectomy are randomly allocated to receive propofol-based TIVA (n=35) or remimazolam-based TIVA (n=35). The recovery profile including the time from the end of anesthetic administration to eye-opening, the time from the end of anesthetic administration to extubation, hemodynamic stability, stability of anesthetic depth, duration of post-anesthetic care stay, the incidence of postoperative nausea and vomiting during the first 24 hours, and the quality of recover 24 hours after surgery using the quality of recovery-15 was assessed by an investigator. The primary outcome is the time from the end of anesthetic administration to eye-opening.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective thyroidectomy under general anesthesia
* American Society of Anesthesiologists (ASA)physical classification I-II
* Willingness and ability to sign an informed consent document

Exclusion Criteria:

* American Society of Anesthesiologists (ASA)physical classification III or more
* BMI > 40kg/m^2
* Allergies to anesthetic or analgesic medications (benzodiazepines, propofol, remifentanil, fentanyl citrate, rocuronium bromide, sugammadex, flumazenil)
* Patients who receive mechanical ventilation morethan 2 hours after surgery
* Patients who receive the following medications within 24 hours prior to general anesthetics: anxiolytics, antipsychotics, rifampicin, succinycholine, neostigmine, flumazenil, cyclosporin
* Patients with galactose intolerance or Lapp Lactase deficiency or glucose-galactose malabsorption
* Medical or psychological disease that can affect the treatment response

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-09-11 (Actual)

PRIMARY OUTCOMES:
Difference in eye opening time between the two groups | Up to the first eye opening from stopping injection of anesthetics
  difference in eye opening time after stopping injection of anesthetics (From the end of anesthetic administration to the first eye opening)

SECONDARY OUTCOMES:
Difference in extubation time between the two groups | Up to extubation from stopping injection of anesthetics
  difference in extubation time after stopping injection of anesthetics (From the end of anesthetic administration to extubation)
Modified Aldrete score | Within 5 minutes of arrival at the post-anesthetic care unit
  Modified Aldrete score (0-10, higher scores mean a better outcome) measured when admit the post-anesthetic care unit
length of post-anesthetic care unit stay | immediately after discharge from the post-anesthetic care unit
  length of post-anesthetic care unit stay (minute)
Postoperative nausea and vomiting during the first 24 hours postoperatively | during the first 24 hours postoperatively
  Incidence of postoperative nausea and vomiting during the first 24 hours postoperatively
postoperative quality of recovery | at 24 hours postoperatively
  quality of recovery measured by the Korean version of the Quality of Recovery-15 (QoR-15K, 0-150, higher scores mean a better outcome)
Intraoperative hemodynamic stability | during the operation
  Intraoperative hemodynamic measured by performance error (%), median performance error (%), median absolute performance error (%), and wobble (%)
Intraoperative anesthetic depth stability | during the operation
  Intraoperative anesthetic depth stability measured by performance error (%), median performance error (%), median absolute performance error (%), and wobble (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Wesolowski AM, Zaccagnino MP, Malapero RJ, Kaye AD, Urman RD. Remimazolam: Pharmacologic Considerations and Clinical Role in Anesthesiology. Pharmacotherapy. 2016 Sep;36(9):1021-7. doi: 10.1002/phar.1806. Epub 2016 Sep 1. PMID 27496519
- [Derived] Lee HJ, Lee HB, Kim YJ, Cho HY, Kim WH, Seo JH. Comparison of the recovery profile of remimazolam with flumazenil and propofol anesthesia for open thyroidectomy. BMC Anesthesiol. 2023 May 2;23(1):147. doi: 10.1186/s12871-023-02104-1. PMID 37131126